CLINICAL TRIAL: NCT05399160
Title: Effect of Nurse-led Supportive Care on Quality of Life in Women With Breast Cancer: An Assessor-blinded, Parallel Group, Randomized Controlled Trial
Brief Title: Effect of Nurse-led Supportive Care on Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Pinar Zorba Bahceli, PhD RN, Asistant Professor, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/270
Record Dates: First submitted 2022-05-24; First posted 2022-06-01 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Quality of Life
Keywords: Nurse-led care; Quality of life; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-led Supportive Care Group (Experimental)
  Interventions: Behavioral: Nurse-led Supportive Care
- Control Group (No Intervention): The control group did not receive any intervention during the study period.

INTERVENTIONS:
Behavioral: Nurse-led Supportive Care — Nurse-led supportive care was given to women who had breast surgery and planned to receive chemotherapy. Nurse-led supportive care was applied to women for eight weeks in the form of face-to-face clinic and telephone interviews.It took an average of 30 minutes to interview women with breast cancer at the clinic, and 15 minutes on average by phone.
  Arms: Nurse-led Supportive Care Group

SUMMARY:
Breast cancer is the most common type of cancer in women with a high mortality rate in the world. The several methods are used in the treatment of breast cancer. One or more of these methods can be preferred according to the characteristics of women with breast cancer. Women may experience many different physiological and psychological symptoms during each treatment process.This situation negatively affects the quality of life of women with breast cancer. For this reason, there is a need for an intervention that could improve quality of life in women with breast cancer. In the literature, it is stated that nurse-led supportive care can be an effective nursing intervention to improve the quality of life in women with breast cancer.

DETAILED DESCRIPTION:
This an assessor-blinded, parallel group randomized controlled trial aimed that investigating the effect of nurse-led supportive care on quality of life in women with breast cancer. This trial was conducted in the general surgery clinic of training and research hospital located in Turkey. All patients were women who had breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older women,
* Stages II or III breast cancer
* Having breast cancer surgery
* Planned to receive chemotherapy
* Able to use a phone
* Who agreed to participate in the study

Exclusion Criteria:

* Having communication problems
* Having psychological diseases
* Receiving any supportive care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life questionnaire-Core Questionnaire (QLQ-C30) | Change from Baseline Quality of Life score at 9th weeks.
  The scale was developed to assess the quality of life of cancer patients. It contains three domains that measure global health status/quality of life, functional and symptom status. Global quality of life is assessed using global health status and quality of life. Functional status consists of the following five subscales: physical function, role function, emotional function, cognitive function and social function. Symptom status consists of the following nine subscales: fatigue, nausea and vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea and financial difficulties. The total score that can be obtained from the scale ranges from 0 to 100. The internal consistency of scale in the Turkish version was determined as 0.90.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Bakircay University Health Sciences Faculty, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yazicioglu Kucuk B, Zorba Bahceli P. The Effects of Nurse-Led Supportive Care Program on Quality of Life in Women with Breast Cancer Receiving Adjuvant Chemotherapy: A Randomized Controlled Pilot Study. Semin Oncol Nurs. 2024 Apr;40(2):151609. doi: 10.1016/j.soncn.2024.151609. Epub 2024 Mar 2. PMID 38433074